CLINICAL TRIAL: NCT06654076
Title: Evaluating Ultra-Sensitive mNGS, Real-Time PCR, Galactomannan, and Lateral-Flow Device for Diagnosing Invasive Fungal Disease in Lung Transplantation: A Retrospective Cross-Sectional Study
Brief Title: Assessing Diagnostic Methods for Invasive Fungal Disease in Lung Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhibin Xu, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: GS001
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Invasive Fungal Disease; Lung Transplant Recipients; Invasive Pulmonary Aspergillosis; Pneumocystis Jirovecii Pneumonia
Keywords: mNGS; Real-time PCR; Galactomannan Assay; Lateral-flow Device; Bronchoalveolar Lavage Fluid; Diagnostic Methods; Lung Transplantation; Fungal Infection
MeSH Terms: conditions — Invasive Fungal Infections; Invasive Pulmonary Aspergillosis; Pneumonia, Pneumocystis; Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The biospecimens used in this study were bronchoalveolar lavage fluid (BALF) samples, collected from lung transplant recipients. These samples were used for diagnostic testing, including metagenomic next-generation sequencing (mNGS), real-time PCR, galactomannan (GM) assay, and lateral-flow device (LFD) tests, to evaluate invasive fungal disease. No DNA retention for future use is applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the diagnostic performance of different tests, including metagenomic next-generation sequencing (mNGS), real-time PCR, galactomannan assay, and lateral-flow device tests, in detecting invasive fungal disease in lung transplant recipients using bronchoalveolar lavage fluid samples. The study is retrospective and cross-sectional in design.

DETAILED DESCRIPTION:
This retrospective, cross-sectional study evaluates the diagnostic accuracy of various tests in detecting invasive fungal disease (IFD) in lung transplant recipients. The diagnostic methods under assessment include metagenomic next-generation sequencing (mNGS), real-time polymerase chain reaction (PCR), galactomannan (GM) assay, and lateral-flow device (LFD) testing, all performed on bronchoalveolar lavage fluid (BALF) samples. The study analyzes the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of each method for diagnosing invasive pulmonary aspergillosis (IPA) and Pneumocystis jirovecii pneumonia (PJP). The sample cohort consists of 109 lung transplant recipients, with data collected from January 2015 to April 2023

ELIGIBILITY:
Inclusion Criteria:

* Adult lung transplant recipients aged 18 years and older.
* Suspected cases of invasive fungal infection (invasive pulmonary aspergillosis or -Pneumocystis jirovecii pneumonia) based on clinical symptoms, radiological findings, or microbiological evidence.
* Able to provide sufficient bronchoalveolar lavage fluid (BALF) samples for diagnostic testing.

Exclusion Criteria:

* Patients with confirmed non-fungal infections.
* Patients unable to provide adequate BALF samples for analysis.
* Patients with severe comorbidities that prevent study participation or completion.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent lung transplantation and were suspected of having invasive fungal infections (IPA or PJP) based on clinical symptoms, radiological findings, or microbiological results. The study includes adults aged 18 and above who were treated at a tertiary hospital from January 2015 to April 2023.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of mNGS for Invasive Pulmonary Aspergillosis and Pneumocystis jirovecii Pneumonia | From January 2015 to April 2023
  Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of metagenomic next-generation sequencing (mNGS) in diagnosing invasive pulmonary aspergillosis (IPA) and Pneumocystis jirovecii pneumonia (PJP) using bronchoalveolar lavage fluid (BALF) samples.

SECONDARY OUTCOMES:
Comparison of Diagnostic Accuracy between mNGS and Other Methods | From January 2015 to April 2023.
  Comparative analysis of diagnostic accuracy, including sensitivity and specificity, between mNGS, real-time PCR, Galactomannan (GM) assay, and lateral-flow device (LFD) tests for detecting IPA and PJP in lung transplant recipients.